CLINICAL TRIAL: NCT02785835
Title: Hepatocellular Carcinoma in HIV-infected Patients
Acronym: GEHEP-002
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Valme (Other)
Responsible Party: Principal Investigator, Nicolás Merchante, MD, PhD, Hospital Universitario de Valme
Other Study IDs: GEHEP-002; RIS-VAC12 (Other: Instituto de Salud Carlos III)
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; HIV; Chronic Hepatitis C; Hepatitis B Virus; Liver Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C, Chronic; Hepatitis B; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study. All HIV-infected patients who have been diagnosed of hepatocellular carcinoma (HCC), following the American Association for the Study of Liver Diseases (AASLD) criteria, in the participant centers are included. Epidemiological, clinical and laboratory data are collected. The clinical and epidemiological characteristics of HCC cases will be analyzed. The efficacy and outcomes after modalities of HCC therapy will be assessed. Mortality and its predictors will be also assessed. In those cases infected by hepatitis C virus (HCV), the impact of HCV therapy on outcomes will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Diagnosis of hepatocellular carcinoma according to American Association for the Study of Liver Diseases (AASLD) criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who are diagnosed of hepatocellular carcinoma following AASLD criteria.
Sampling Method: Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2014-05; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | At 1 year
  Overall survival after HCC diagnosis at 1 year

CONTACTS AND LOCATIONS:
Locations (30):
- Spain (30):
  - Hospital de Orihuela, Orihuela, Alicante
  - Hospital Clínico Universitario de San Juan, Sant Joan d'Alacant, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital German Trias i Pujol, Badalona, Barcelona
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital de La Linea, La Línea de la Concepción, Cádiz
  - Hospital Universitario de Donostia, San Sebastián, Guipúzcua
  - Hospital Universitario A Coruña, A Coruña, La Coruña
  - Hospital de San Pedro, Logroño, La Rioja
  - Hospital de Santa Lucía, Cartagena, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de San Eloy, Barakaldo, Vizcaya
  - Hospital de Basurto, Basurto, Vizcaya
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Puerto Real, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario de Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario La Princesa, Madrid
  - Hospital Regional Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Arrixaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Merchante N, Merino E, Rodriguez-Arrondo F, Tural C, Munoz J, Delgado-Fernandez M, Jover F, Galindo MJ, Rivero A, Lopez-Aldeguer J, Aguirrebengoa K, Romero-Palacios A, Martinez E, Pineda JA. HIV/hepatitis C virus-coinfected patients who achieved sustained virological response are still at risk of developing hepatocellular carcinoma. AIDS. 2014 Jan 2;28(1):41-7. doi: 10.1097/QAD.0000000000000005. PMID 24056067
- [Result] Merchante N, Merino E, Lopez-Aldeguer J, Jover F, Delgado-Fernandez M, Galindo MJ, Ortega E, Rivero A, Minguez C, Romero-Palacios A, Padilla S, Marquez-Solero M, Amador C, Rios-Villegas MJ, Tellez F, Portilla J, Pineda JA. Increasing incidence of hepatocellular carcinoma in HIV-infected patients in Spain. Clin Infect Dis. 2013 Jan;56(1):143-50. doi: 10.1093/cid/cis777. Epub 2012 Sep 5. PMID 22955438
- [Result] Merchante N, Ibarra S, Revollo B, Rodriguez-Arrondo F, Merino E, Delgado-Fernandez M, Montero-Alonso M, Tellez F, Galindo MJ, Rivero-Juarez A, Garcia MA, Minguez C, Romero-Palacios A, Garcia-Deltoro M, Pineda JA; GEHEP-002 Study Group. Real-life experience with sorafenib for the treatment of hepatocellular carcinoma in HIV-infected patients. AIDS. 2017 Jan 2;31(1):89-95. doi: 10.1097/QAD.0000000000001293. PMID 27755109
- [Result] Merchante N, Rodriguez-Arrondo F, Revollo B, Merino E, Ibarra S, Galindo MJ, Montero M, Garcia-Deltoro M, Rivero-Juarez A, Tellez F, Delgado-Fernandez M, Rios-Villegas MJ, Garcia MA, Vera-Mendez FJ, Ojeda-Burgos G, Lopez-Ruz MA, Metola L, Omar M, Aleman-Valls MR, Aguirrebengoa K, Portu J, Raffo M, Macias J, Pineda JA; GEHEP-002 Study Group. Hepatocellular carcinoma after sustained virological response with interferon-free regimens in HIV/hepatitis C virus-coinfected patients. AIDS. 2018 Jul 17;32(11):1423-1430. doi: 10.1097/QAD.0000000000001809. PMID 29596108
- [Result] Pinato DJ, Allara E, Chen TY, Trevisani F, Minguez B, Zoli M, Harris M, Dalla Pria A, Merchante N, Platt H, Jain M, Caturelli E, Kikuchi L, Pineda J, Nelson M, Farinati F, Rapaccini GL, Aytaman A, Yin M, Tan CK, Bower M, Giannini EG, Brau N; Liver Cancer in HIV and ITA.LI.CA Study Groups. Influence of HIV Infection on the Natural History of Hepatocellular Carcinoma: Results From a Global Multicohort Study. J Clin Oncol. 2019 Feb 1;37(4):296-304. doi: 10.1200/JCO.18.00885. Epub 2018 Dec 18. PMID 30562130
- [Result] Merchante N, Figueruela B, Rodriguez-Fernandez M, Rodriguez-Arrondo F, Revollo B, Ibarra S, Galindo MJ, Merino E, Montero M, Tellez F, Garcia-Deltoro M, Rivero-Juarez A, Delgado-Fernandez M, Rios-Villegas MJ, Aguirrebengoa K, Garcia MA, Portu J, Vera-Mendez FJ, Villalobos M, Minguez C, De Los Santos I, Lopez-Ruz MA, Omar M, Galera C, Macias J, Pineda JA; GEHEP-002 Study Group. Low performance of ultrasound surveillance for the diagnosis of hepatocellular carcinoma in HIV-infected patients. AIDS. 2019 Feb 1;33(2):269-278. doi: 10.1097/QAD.0000000000002065. PMID 30325782